CLINICAL TRIAL: NCT06159491
Title: Pacritinib in Combination With Azacitidine in Patients With Chronic Myelomonocytic Leukemia
Brief Title: Pacritinib in CMML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Douglas Tremblay (Other)
Collaborators: Sobi, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Douglas Tremblay, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 23-1514
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Azacitidine

STUDY DESIGN:
Intervention Model Description: Phase I will follow a 3+3 design in phase I with starting dose of 200mg with possibility of de-escalation if more than 1/3 or 1/6 experience DLT. Phase I will require 6-12 patients to select the MTD.
  Phase II, if MTD selected in Phase I, will follow a Simon's two stage design. The null hypothesis that the true response rate is 55% will be tested against a one-sided alternative that the response rate is 80%. In the first stage, 6 patients treated at the MTD from Phase I will be included. If there are 3 or fewer responses in these 6 patients, the study may be stopped. Otherwise, 12 additional patients will be accrued for a total of 18. The null hypothesis will be rejected if 13 or more responses are observed in 18 patients. This design yields a type I error rate of 9% and power of 82% when the true response rate is 80%.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pacritinib in combination with Azacitidine (Experimental): Participants will take pacritinib 200 mg BID for each 28 day cycle, azacitidine 75mg/m2 will be administered IV or SQ QD D1-7 of each 28 day cycle
  Interventions: Drug: Pacritinib; Drug: Azacitidine

INTERVENTIONS:
Drug: Pacritinib — Participants will take Pacritinib 100 mg - 200mg BID for each 28 day cycle
Drug: Azacitidine — Azacitidine 75mg/m^2 will be administered IV or SQ QD D1-7 of each 28 day cycle

SUMMARY:
This is a phase 1/2 trial of pacritinib in combination with azacitidine in patients with Chronic Myelomonocytic Leukemia (CMML). Patients will be newly diagnosed or previously treated but could not have received a prior JAK inhibitor. Patients who have previously been treated with a hypomethylating agent (HMA) must have received ≤ 1 cycle. Pacritinib will be initially tested at a dose of 200mg twice daily (dose level 0) in combination with azacitidine 75mg/m2, which can be administered subcutaneously or intravenously, for 7 days in a 28-day cycle. If there are 2 DLTs in the first 6 patients, there will be a dose escalation to pacritinib 100mg twice daily (dose level -1) and an additional 6 patients will be enrolled. Based on the phase 1, 3+3 dose de-escalation design, 6-12 patients will be enrolled in the phase 1 portion. After the completion of phase 1 and identification of the recommended phase 2 dose (RP2D), the trial will then proceed to phase 2 which will employ a Simon two stage design. This portion will include the 6 patients enrolled during the phase 1 portion at the MTD. An interim analysis for futility will occur. If 3 or fewer patients have had a clinical benefit (CB) or better, as defined by 2015 MDS/MPN IWG criteria, the PI and DSMC will meet to discuss the totality of the evidence and determine if the trial shall proceed. In the second stage, an additional 12 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age at time of signing the Informed Consent Form (ICF).
* Participants must voluntarily sign an ICF.
* Participants must have a pathologically confirmed diagnosis of chronic myelomonocytic leukemia per World Health Organization (WHO) or International Consensus Classification (ICC)
* Participants must be JAK inhibitor naïve.
* Participants may be hypomethylating agent (HMA) naïve or can be treated with up to one prior cycle.
* Participants must have either proliferative CMML (WBC ≥13 x 109/L) or have intermediate-2 or high risk CMML by the clinical/molecular CMML-specific prognostic scoring system (CPSS-Mol).
* Participants must have a life expectancy of at least 24 weeks per investigator.
* ECOG performance status ≤ 3.
* Females of reproductive potential should use effective contraception during treatment with azacitidine and for 6 months after the last dose and males with female partners of reproductive potential should use effective contraception during treatment with azacitidine and for 3 months after the last dose.
* Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy.
* Must have adequate organ function as demonstrated by the following:

  * Serum total bilirubin ≤ 2.0 x upper limit of normal (ULN) unless considered due to leukemic organ involvement, Gilbert's syndrome, or hemolysis.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN.
  * Creatinine clearance (CrCl) of ≥30 mL/min.
  * PT or INR <=1.5x ULN and PTT or aPTT <=1.5x ULN.
  * ANC >= 500 cells/μL.
* Ability to adhere to the study visit schedule and all protocol requirements.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 2 weeks or within 5 half-lives of the prior investigational agent, whichever is shorter, of the first dose of treatment.
* Active Graft Versus Host Disease (GVHD), or any GVHD requiring treatment with immunosuppression, with the exception of topical steroids and systemic steroids at a dose equivalent to prednisone 10mg or less and at a stable or decreasing dose. Any GVHD treatment (including calcineurin inhibitors) must be discontinued at least 28 days prior to Day 1 of study treatment.
* Systemic treatment with a strong CYP3A4 inhibitor or a strong CYP450 inducer within 14 days prior to treatment Day 1 (see Appendix 13.7 and 13.8 for a list of CYP3A4 inhibitors and CYP450 inducers, respectively). Shorter washout periods may be permitted with approval of the Study Chair, provided that the washout period is at least five half-lives of the drug prior to treatment Day 1.
* Other invasive malignancies within the last 3 years, except curatively treated non-melanoma skin cancer, localized prostate, cervical cancer, and any curatively treated carcinoma in situ.
* Presence of active serious infection.

  * If a patient is identified to have COVID-19 during the screening period, participants may be considered eligible if in the opinion of the investigator there are no COVID-19 sequlae that may place the patient at a higher risk of receiving investigational treatment.
* Any serious, unstable medical or psychiatric condition that would prevent, (as judged by the Investigator) the patient from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Known history of uncontrolled human immunodeficiency virus (HIV).
* Significant recent bleeding history defined as NCI CTCAE grade ≥2 within 3 months prior to treatment Day 1, unless precipitated by an inciting event (e.g., surgery, trauma, or injury).
* Systemic treatment with medications that increase the risk of bleeding, including anticoagulants, antiplatelet agents (except for aspirin dosages of ≤100 mg per day), anti-vascular endothelial growth factor (anti-VEGF) agents, and daily use of COX-1 inhibiting Non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to treatment Day 1.
* Any history of CTCAE grade ≥2 cardiac conditions within 6 months prior to treatment Day 1. Patients with asymptomatic grade 2 non-dysrhythmia cardiovascular conditions may be considered for inclusion, with the approval of the Study Chair, if stable and unlikely to affect patient safety.
* Heart failure other than NYHA class I (asymptomatic, without limitation).
* QT corrected by the Fridericia method (QTcF) prolongation >480 ms or other factors that increase the risk for QT interval prolongation (e.g., hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or history of long QT interval syndrome).
* Known active systemic hepatitis B, or C infection requiring therapy or known cirrhosis.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or pharmaceutical sponsor staff directly involved with this trial, unless prospective IRB approval (by chair or designee) is given allowing exception to this criterion for a specific participant.
* Organ transplant recipients other than bone marrow transplant.
* Women who are pregnant or lactating.
* Patient with known gastrointestinal (GI) disease or prior GI procedure that could interfere with the oral absorption or tolerance of pacritinib, including difficulty swallowing, are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity of Pacritinib in combination with Azacitidine | at the end of one 28-day cycle
  Phase 1: The recommended phase 2 dose (RP2D) for the combination of pacritinib with azacitidine will be determined based on the dose limiting toxicity (DLT) rate, defined as the proportion of participants in the DLT-evaluable population that experience a DLT within the first 4 weeks (1 cycle) of initiating treatment at the recommended phase 2 dose.
Proportion of participants that achieve clinical benefit or better measured using 2015 MDS/MPN IWG Criteria | 24 weeks (6 cycles, each cycle is 28 days)
  Phase 2: The preliminary efficacy of pacritinib in combination with azacitidine will be defined as the proportion of participants that achieve clinical benefit or better within 24 weeks (6 cycles, each cyce) of initiating treatment. Clinical benefit as defined by 2015 MDS/MPN IWG criteria within erythroid response, platelet response, neutrophil response, spleen response or symptom response.
Overall Response Rate (ORR) to measure clinical benefit | 24 weeks (6 cycles, each cycle is 28 days)
  Clinical benefit will be determined by evaluating overall response rate (ORR) which is defined by complete remission.

SECONDARY OUTCOMES:
Number of Adverse events Grade 3 or higher measured using NCI CTCAE Version 5.0 | up to 30 days after last study dose (up to 6 cycles, each cycle 28 days)
  Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE Version 5.0. Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.
Duration of Response (DOR) to measure efficacy | up to 24 months
  Preliminary efficacy of the combination of pacritinib with azacitidine as determined by duration of response (DOR). DOR is the length of time that a tumor continues to respond to treatment without the cancer growing or spreading.
Overall Survival (OS) to measure efficacy | up to 24 months
  Preliminary efficacy of the combination of pacritinib with azacitidine as determined by duration of overall survival (OS). OS is defined as the time from the first dose of study treatment to the date of death (whatever the cause).
Disease Free Survival (DFS) to measure efficacy | up to 24 months
  Preliminary efficacy of the combination of pacritinib with azacitidine as determined by disease free survival (DFS). DFS is defined as the time from randomization to recurrence of tumor or death.
Change in Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SASF TSS) | Baseline and after 3 and 6 cycles of therapy, each cycle is 28 days
  Change in MPN-SAF TSS to determine differences in health-related quality of life before and after treatment. MPN-SAF TSS has a possible range of 0-100, with higher score indicating higher level of symptom severity.
Percentage of patients achieving "very much" or "much" in the Patient Global Impression of Change (PGIC) | Baseline and after 3 and 6 cycles of therapy, each cycle is 28 days
  Patient Global Impression of Change (PGIC) to determine differences in health-related quality of life before and after treatment. Percentage of patients achieving "very much" or "much" improved as measured by Patient Global Impression of Change (PGIC) will be recorded. The Patient's Global Impression of Change (PGIC) will be used to assess self-reported relieving effect. It will evaluate pain from no change (score 0-1), minimally improved (score 2-3), much improved (score 4-5), and very much improved (score 6-7). Full score from 0-7, with higher score indicating more improvement.
Change in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | Baseline and after 3 and 6 cycles of therapy, each cycle is 28 days
  Change in EORTC-QLQ-C30 score to determine differences in health-related quality of life before and after treatment. EORTC QLC-C30 is a 30-item questionnaire to assess the quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); two used 7-point scale (1 'Very Poor' to 7 'Excellent'). Subscales and Total Scale are averaged, and transformed to 0-100 scale; with higher score indicating better quality of life
Change in Palpable Spleen Size | Baseline and after 3 and 6 cycles of therapy, each cycle is 28 days
  Change in palpable spleen size to determine differences in health-related quality of life before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Tremblay, MD, Principal Investigator — Icahn School of Medicine
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Specify Other Mechanism Request submitted to Principal Investigator via e-mail: douglas.tremblay@mssm.edu.